CLINICAL TRIAL: NCT03200808
Title: Evaluation of the Efficacy of Mixed Methylene Blue Compound Injection for the Treatment of Nonneoplastic Epithelial Disorders of Vulva.
Brief Title: Methylene Blue Injection for Nonneoplastic Epithelial Disorders of Vulva
Acronym: NNEDsMB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maternal and Child Health Hospital of Hubei Province (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NNEDs
Record Dates: First submitted 2017-06-25; First posted 2017-06-27 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Nonneoplastic Epithelial Disorders of Vulva
Keywords: Nonneoplastic Epithelial Disorders; methylene blue; treatment

STUDY DESIGN:
Intervention Model Description: Pations with nonneoplastic epithelial disorders（NNEDS） of vulva.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment group (Experimental): Methylene blue compound injection are mixed by Methylene Blue injection, Dexamethasone powder-injection, Ropivacaine injection and Normal saline injection. Each individual component can help in a very wide range of medical conditions without serious side effects.
  Every patient received intradermal mixed methylene blue compound injection twice. All patients were observed during the hospitalization at the first injection, and two weeks later they received the second injection at the outpatient department.
  Interventions: Drug: mixed methylene blue compound injection

INTERVENTIONS:
Drug: mixed methylene blue compound injection — Every patient received intradermal mixed methylene blue compound injection twice.

SUMMARY:
The aim of this study is to demonstrate the safety and effectiveness of mixed methylene blue compound Injection for the treatment of nonneoplastic epithelial disorders（NNEDS） of vulva.

NNEDS of skin and mucosa of vulva refer to a group of chronic diseases including squamous hyperplasia and lichen sclerosus, which mainly cause vulvar itching and hypopigmentation. Usually the itching is severe may influence social activities and sleep. In addition, NNEDS cause scarring of the vulva which may cause significant sexual dysfunction or pain. The reasons for NNEDs are not clear and the methods of treatment are diverse. The current treatments are primarily local drug (e.g. steroid, calcineurin inhibitors, immunosuppressive agents ), surgical treatments, laser or photodynamic therapy, and the "gold standard" treatment for lichen sclerosus is potent steroids creams. However, all the treatments are not good enough, and the diseases often recur and severely affect women's quality of life. So the investigators reviewed plenty of literatures, and found some authors used single intradermal 1% methylene blue injection for intractable idiopathic pruritus ani and the effect was good. As a preliminary experiment, the investigators used intradermal mixed methylene blue compound injection for a NNEDs patient in the year of 2012, the itching of the patient stopped immediately and the color of the vulva recovered 6 months later. The patient keeps healthy till now. And from then on, the investigators designed this study and to verify the effect and complications of intradermal mixed methylene blue compound injection for the treatment of NNEDS. So far, there is no similar study reported internationally.

DETAILED DESCRIPTION:
Methylene blue compound injection are mixed by Methylene Blue injection, Dexamethasone powder-injection, Ropivacaine injection and Normal saline injection. Each individual component can help in a very wide range of medical conditions without serious side effects.

In this study，the investigators used methylene blue compound injection intradermally to treat NNEDs patients. Patients with a diagnosis of biopsy proven NNEDs from Maternal and Child Health Hospital of Hubei Province (China) between October 2013 to October 2016 were recruited. Every patient received intradermal mixed methylene blue compound injection twice. All patients were observed during the hospitalization at the first injection, and two weeks later they received the second injection at the outpatient department. Ages, itching scores, percentage of hypopigmented skin, and recurrences were recorded through inquiry and physical examination before and after treatment. Side effects (such as edema, fever and vulva pain) were also recorded. All women were followed up 1, 3, 6, 12 months after treatment, which included inquiry and physical examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically and biopsy confirmed non-neoplasia epithelial disorders of skin and mucosa of vulva.
* Patient must have a score of 5 or greater in the itching score table before treatment and the itching must last at least 6 months.

Exclusion Criteria:

* Patients with vulvovaginal or other gynecological trauma, acute inflammatory diseases and other acute illness
* Patients have been treated with any kind of topical therapy at the vulva within 12 weeks prior to participation in the study
* Patients with other serious diseases (e.g. liver or kidney diseases) that need immediate treatment
* Patients with atypical vulvar hyperplasia or vulvar cancer confirmed by biopsy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
itching scores | 1 years
  The patients rate the itching on a visual analogue scale (VAS) before and after the treatment. A VAS is a 100-mm long horizontal line with verbal descriptors at each end to express the extremes of the itching feeling. The most severe itching equals to score 10, and no itching equals to score 0. Patients marked the point on the line that best corresponded to their itching severity.

SECONDARY OUTCOMES:
percentage of hypopigmented skin | 1 years
  Doctors rate the hypopigmented skin on a vulva surface area scale (VSAS) before and after treatment through colposcopy. The vulva area is divided into six regions as labia majora, labia minora, interlabial sulci, clitoris and clitoral hood, perineum, and perianal area. The investigators estimated that the area percentage of labia majora, labia minora, interlabial sulci, clitoris and clitoral hood, perineum, and perianal area was 48%, 24%, 4%, 4%, 10% and 10% differently. Among the six regions, interlabial sulci, clitoris and clitoral hood, perineum, and perianal area could be divided into four equal proportions at most when the area percentage was calculated. And each side of labia majora and labia minora could be divided into four equal proportions at most. If all the vulva area is involved, the VSAS score is 100%, and if no area of vulva is involed, the VSAS score is 0%.

OTHER OUTCOMES:
pathology changes | 1 years
  changes of nonneoplastic epithelial disorders from biopsy pathology

CONTACTS AND LOCATIONS:
Overall Officials: Han Gao, bachelor, Study Director — Maternal and Child health Hospital of Hubei Province,Wuhan,China; Xufeng Wu, PH.D, Study Chair — Maternal and Child health Hospital of Hubei Province,Wuhan,China; Yanli Li, Master, Principal Investigator — Maternal and Child health Hospital of Hubei Province,Wuhan,China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neill SM, Lewis FM, Tatnall FM, Cox NH; British Association of Dermatologists. British Association of Dermatologists' guidelines for the management of lichen sclerosus 2010. Br J Dermatol. 2010 Oct;163(4):672-82. doi: 10.1111/j.1365-2133.2010.09997.x. No abstract available. PMID 20854400
- [Background] Samalavicius NE, Poskus T, Gupta RK, Lunevicius R. Long-term results of single intradermal 1 % methylene blue injection for intractable idiopathic pruritus ani: a prospective study. Tech Coloproctol. 2012 Aug;16(4):295-9. doi: 10.1007/s10151-012-0846-1. Epub 2012 Jun 6. PMID 22669483
- [Derived] Li Y, Shi J, Tan W, Ma Q, Wu X, Gao H. Prospective observational study of the efficacy of mixed methylene blue compound injection for treatment of vulvar non-neoplastic epithelial disorders. Int J Gynaecol Obstet. 2020 Feb;148(2):157-161. doi: 10.1002/ijgo.13007. Epub 2019 Nov 19. PMID 31628667